CLINICAL TRIAL: NCT02070848
Title: Muscle Blood Flow Control During Exercise in Humans: Contribution From Mechanical and Metabolic Signals and Role of the Erythrocyte.
Brief Title: Muscle Blood Flow During Exercise
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5456
Record Dates: First submitted 2014-02-14; First posted 2014-02-25 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Skeletal Muscle Blood Flow
Keywords: red blood cell; knee extension exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Concentric vs eccentric: One arm study in which each subject will act as his own control.
  Interventions: Other: Session 1-4; Other: Session 4; Other: Session 5

INTERVENTIONS:
Other: Session 1-4 — Familiarization sessions to knee-extensor exercise separated by 72h recovery
Other: Session 4 — After the last familiarization session, 1 maximal incremental test on a bicycle, followed by 72h rest
Other: Session 5 — 2 maximal incremental tests of knee-extension exercise (concentric vs eccentric), separated by 3h rest.

SUMMARY:
Physical exercise triggers various physiological responses including a marked increase in muscle blood flow and oxygen delivery in order to support muscle activity. How muscle blood flow is controlled is currently unclear.

The primary purpose of this study is to establish the respective contribution of metabolic (linked to energy requirements) and mechanical (linked to muscle tensions) signals in the exercise hyperemia and the possible role of the red blood cells.

Vasodilation and muscle blood flow during exercise are controlled by ATP released in the plasma from the red blood cells in response to a combination of metabolic and mechanical signals applied on the vasculature.

ELIGIBILITY:
Inclusion Criteria:

* Non smoker or having stopped smoking for at least 5 yr
* Practice sports: physical activity level will be evaluated with a questionnaire (de Baecke et coll., 1982) and will give an activity index greater than 6 together with a VO2max greater than 50 ml/kg/min
* Body mass index lower than 25
* Registered to the French Social Security system
* Providing a written and informed consent to participate in the study

Exclusion Criteria:

* History of venous or arterial thrombo-embolic events
* Bad perfusion from the cubital artery
* Unable to understand the information notice
* Subject exposed to law investigations or with financial dependancy
* Subjects feeling unwell whan seing blood.
* Subjects advised to not practice sport.
* Musculo-tendinous or articular issues with the lower leg
* Respiratory, cardiovascular or metabolic pathologies
* Current medical treatment that can not be stopped 7 days before the experiment.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be students recruited in the Faculty, sports clubs...
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Change in leg blood flow during concentric and eccentric muscle work | Leg blood flow measurements during exercises performed at the beginning, after 14 minutes, then after 18 min, 22 min, 26 min, 30 min, 33 min, 35 min and 45 min
  Serial measures (9) of leg blood flow during concentric and eccentric muscle work are performed at the beginning of the exercise (t0), and then after 14 minutes (t14), after 18 minutes (t18), after 22 minutes (t22), after 26 minutes (t26), after 30 minutes (t30), after 33 minutes (t33), after 35 minutes (t35), and after 45 minutes (45) during each exercice, concentric and eccentric.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane DOUTRELEAU, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg; DUFOUR Stéphane, MD, Study Director — Faculté des Sciences du Sport 14 Rue René Descartes 67084 Strasbourg; FAVRET Fabrice, MD, Study Chair — Faculté des Sciences du Sport 14 Rue René Descartes 67084 Strasbourg; LONSDORFER Evelyne, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- SERVICE DE PHYSIOLOGIE ET D'EXPLORATIONS FONCTIONNELLES - Nouvel Hôpital Civil, Strasbourg, France